CLINICAL TRIAL: NCT05787262
Title: Clinical Utility of Upper Endoscopy in Diagnosis of Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Walaa Mohamed Omar, resident at tropical medicine department, sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-03-17MS
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: upper endoscopy — Upper endoscopy , biopsy and histopathological examination of taken biopsies.

SUMMARY:
Helicobacter pylori (H. pylori) is a gram-negative flagellated bacterium that inhabits the gastric environment of 60.3% of the world population, and its prevalence is particularly high in countries with inferior socioeconomic conditions, exceeding 80% in some regions of the globe , This phenomenon occurs among other reasons, due to the unsatisfactory basic sanitation and high people aggregations observed in many under developed nations, scenarios that favour the oral-oral and fecal-oral transmissions of H.pylori.Another possible transmission route of this pathogen is the sexual route.

Several studies have shown that the colonization of H.pylori could be negatively and positively associated with the induction and progression of several diseases .It has been reported to be linked to gastric and duodenal ulcer, gastric carcinoma, and gastric mucosa-associated lymphoid tissue (MALT) lymphoma and gastritis ,A positive association also reported between H.pylori infection and oesophageal cancer.

Moreover, evidence is also available on the positive association between H.pylori and non gastrointestinal diseases such as diabetes mellitus , coronary artery disease

, and anaemia. Abdominal pain and discomfort, nausea, burping, and loss of appetite are common symptoms of H.pylori infection. Other symptoms include, bloating, weight loss, and heart burn.

Several approaches are used in the detection of H. pylori. Both the invasive and the non-invasive methods are employed in the detection of H. pylori in a patient. Many factors, however, influence choices in the method of diagnosis: availability of diagnostic instruments/materials, sampling population, and competency and experience of the physicians/clinicians .

Invasive methods include endoscopic evaluation, histology, rapid urease test (RUT), and bacterial culture. Non-invasive methods include urea breath test (UBT), stool antigen test (SAT), serology, and molecular diagnostic approaches .Endoscopy is an accurate test for diagnosing the infection as well as the inflammation.

Endoscopy also allows the determination of the severity of gastritis with biopsies as well as the presence of ulcers, MALT lymphoma and cancer.

Real-time endoscopy along with conventional white light imaging (WLI)and image enhanced endoscopic (IEE)techniques, such as narrow-band imaging (NBI), linked color imaging (LCI) and blue laser imaging (BLI), appear to have important roles in clinical practice to identify H. pyloriinfected status .

Another endoscopic technique is i-scan digital chromoendoscopy, which is a digital contrast method that enhances minute mucosal structures and subtle changes in color . The overall diagnostic accuracy of i-scan is 97% compared to 78% for WLI .

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) of both genders.
* Symptoms should be present within three months and have started ≥ six months before diagnosis of dyspepsia according to RomeIII criteria.

Exclusion Criteria:

* Previous H.pylori eradication therapy.
* History of gastric surgery.
* Patients declining to provide informed consent.
* Pregnant and lactating women.
* Severe coagulopathy.
* liver cirrhosis, portal hypertensive gastropathy.
* Other causes of chronic gastritis (bile reflux gastritis, Crohn's disease, autoimmune gastritis, chemical gastritis, eosinophilic gastritis).
* Patients without endoscopic features or signs of gastritis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 345 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of cases with H.pylori infection among all patients subjected to upper endoscopy. | 18 months
  Evaluate the diagnostic accuracy of I-scan technique in doagnosis of H.pylori infection

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Chen TP, Hung HF, Chen MK, Lai HH, Hsu WF, Huang KC, Yang KC. Helicobacter Pylori Infection is Positively Associated with Metabolic Syndrome in Taiwanese Adults: a Cross-Sectional Study. Helicobacter. 2015 Jun;20(3):184-91. doi: 10.1111/hel.12190. Epub 2015 Jan 12. PMID 25582223
- [Background] Coelho LGV, Marinho JR, Genta R, Ribeiro LT, Passos MDCF, Zaterka S, Assumpcao PP, Barbosa AJA, Barbuti R, Braga LL, Breyer H, Carvalhaes A, Chinzon D, Cury M, Domingues G, Jorge JL, Maguilnik I, Marinho FP, Moraes-Filho JP, Parente JML, Paula-E-Silva CM, Pedrazzoli-Junior J, Ramos AFP, Seidler H, Spinelli JN, Zir JV. IVTH BRAZILIAN CONSENSUS CONFERENCE ON HELICOBACTER PYLORI INFECTION. Arq Gastroenterol. 2018 Apr-Jun;55(2):97-121. doi: 10.1590/S0004-2803.201800000-20. Epub 2018 Apr 16. PMID 30043876
- [Background] Crowe SE. Helicobacter pylori Infection. N Engl J Med. 2019 Mar 21;380(12):1158-1165. doi: 10.1056/NEJMcp1710945. No abstract available. PMID 30893536
- [Background] Diaconu S, Predescu A, Moldoveanu A, Pop CS, Fierbinteanu-Braticevici C. Helicobacter pylori infection: old and new. J Med Life. 2017 Apr-Jun;10(2):112-117. PMID 28616085